CLINICAL TRIAL: NCT02307734
Title: A Family-Focused Intervention for Asian American Male Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of California, Davis (Other); Chinese Community Health Resource Center (Other); Immigrant Resettlement & Cultural Center (Unknown); Vietnamese Voluntary Foundation, Inc. (Other); Southeast Asian Community Center (Unknown); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01DA036749 (NIH); R01DA036749 (NIH)
Record Dates: First submitted 2014-11-24; First posted 2014-12-04 (Estimated); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Smoking Cessation; Family; Health Behavior
Keywords: Lay Health Workers; Chinese; Vietnamese; Tobacco Use; Intervention; Behavior Change; Social Networks; Asians
MeSH Terms: conditions — Smoking Cessation; Health Behavior; Tobacco Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Quit Smoking for a Healthy Family (Experimental): The experimental/intervention study arm focuses on providing smoking cessation education and support through 2 LHW outreach small group educational sessions (4-5 weeks apart) and 2 individual follow-up telephone calls to smoker and family participants separately.
  Interventions: Behavioral: Quit Smoking for a Healthy Family
- Healthy Living (Active Comparator): In this comparison arm, participants will receive the same number of contacts on the same schedule and in the same format (2 small group sessions and 2 telephone calls). The comparison LHWs will receive training about "Healthy Living" focusing on nutrition and physical activity education. Participants will also receive the Smoking Cessation Resource Handout.
  Interventions: Behavioral: Healthy Living

INTERVENTIONS:
Behavioral: Quit Smoking for a Healthy Family — The experimental/intervention study arm focuses on providing smoking cessation education and support through 2 LHW outreach small group educational sessions (4-5 weeks apart) and 2 individual follow-up telephone calls to smoker and family participants separately at 2-3 weeks after each group session for a total of 4 intervention contacts over 2 months. The LHW and dyads will choose the site of sessions, such as the LHW's or a participant's home, or LHW Agency's office. Each small group session will last 90 minutes, be interactive, and involve sharing personal stories, learning using a flip chart, and setting individual goals. Each telephone call will be 15- 20 minutes to reinforce progress and provide support.
  Arms: Quit Smoking for a Healthy Family
Behavioral: Healthy Living — In this comparison arm, participants will receive the same number of contacts on the same schedule and in the same format (2 small group sessions and 2 telephone calls). The comparison LHWs will receive training about "Healthy Living" focusing on nutrition and physical activity education. Participants will also receive the Smoking Cessation Resource Handout.
  Arms: Healthy Living

SUMMARY:
This project proposes two aims. The first aim is to evaluate the efficacy of a family-focused intervention in promoting smoking cessation in Chinese and Vietnamese male smokers using a 2-arm cluster randomized controlled trial with assessments at baseline, 6, and 12 months targeting 360 smoker-family dyads. Half of the participants will be assigned to the proposed intervention, and the remaining half will be assigned to an attention-control condition where they will receive education on healthy eating and physical activity. The second aim is to explore mediators to identify key psychosocial and behavioral processes that underlie how the intervention affects the processes of quitting and maintaining abstinence in Chinese and Vietnamese smokers.

DETAILED DESCRIPTION:
Smoking prevalence remains high in subgroups of Asian American men, particularly among those with low English proficiency (LEP) and immigrants from cultures where smoking prevalence is high, including Chinese and Vietnamese. The 2011-12 California Health Interview Survey estimates that nearly half (46%) of all Asian male smokers in California are either Chinese or Vietnamese. The smoking prevalences among LEP Chinese and Vietnamese men were 32% and 43%, respectively, compared to 16% of the general California male population. The investigators developed a family-focused intervention utilizing lay health worker (LWH) outreach that integrates formative qualitative research and selected constructs from Social Network Theory, Social Cognitive Theory, and the Transtheoretical Model. The intervention involves 2 small group education sessions with dyads of smokers and family members, and 2 follow-up individual telephone calls delivered by LHWs over 2 months. Our single-group pilot trial with 96 dyads of Chinese and Vietnamese male daily smokers and their family members showed a high feasibility of recruiting unmotivated smokers (42% were at "precontemplation"), and a promising 7-day point prevalence abstinence rate of 30% at 3 months with independent corroboration from family members. The first aim of the study is to evaluate the efficacy of the family-focused intervention in promoting smoking cessation in Chinese and Vietnamese male smokers. The second aim is to explore mediators to identify key psychosocial and behavioral processes that underlie how the intervention affects the processes of quitting and maintaining abstinence. The investigators will conduct a 2-arm cluster randomized controlled trial (RCT) with assessments at baseline, 6 and 12 months following intervention initiation. The RCT involves 60 lay health workers (LHWs); each recruits and delivers interventions to 6 dyads of one male daily smoker and one family member from his household, for a total 360 smoker-family dyads. Half of the LHWs, stratified by Asian subgroup and smoking history, will be randomized to the family-focused intervention group and the other half will be assigned to an attention control condition receiving education on healthy eating. All participants will receive written information on smoking cessation resources. The investigators hypothesize that, at 6 and 12 month follow-up, the intervention smokers will be more likely to achieve biochemically verified smoking abstinence (7-day point prevalence), to report having made at least one 24-hour quit attempt, and to report using at least one evidence-based smoking cessation resource (telephone counseling or Quitline, medication, health professional advice) than smokers in the control condition. Using prospective quantitative data obtained from the RCT, and post-trial dyadic and individual interviews of 12 smokers and 12 family members selected based on abstinence experiences, the investigators will explore mediators at individual, family and social network levels that explain how the intervention affects quitting and maintaining abstinence. The long-term goal is to understand effective ways to utilize family-based and social outreach strategies to reduce tobacco use disparities in hard-to-reach populations.

ELIGIBILITY:
Inclusion Criteria (for smoker participants):

* Chinese or Vietnamese males
* Age > 18
* Speak Cantonese or Mandarin (major Chinese dialects) or Vietnamese
* Have smoked at least 1 cigarette daily during the past 7 days, have a family member in the household with whom he will participate in the study, plan to stay in the area for the next 3 months (to complete all intervention activities) and can provide a valid phone number and a mailing address (for follow-up assessments and for sending saliva sample collection kits and payments).

Exclusion Criteria (for smoker participants):

* Those who are currently in a smoking cessation program or trying to quit smoking with assistance will be excluded.

Inclusion Criteria (for family participants):

* Family members (male or female) of an eligible smoker
* Age > 18
* Speak Cantonese or Mandarin (major Chinese dialects) or Vietnamese
* Have never smoked or have formerly smoked but have not had any cigarette in the year prior to participation

Exclusion Criteria (for family participants):

* Only one smoker-family dyad from a household may participate.
* They must not live in the same household as their own LHW (or another LHW) or have participated in the study at any time (e.g., focus groups not directly related to the intervention implementation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 680 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
long-term 7-day point prevalence smoking abstinence (smoker participants) | 12 months
  Salivary cotinine will be obtained to provide biochemical verification for participants who report abstinence. A cotinine level of < 12 ng/mL will be considered to verify abstinence. Since nicotine replacement therapy (NRT) use will also produce positive cotinine assays, for participants reporting concurrent NRT use, we will use independent corroboration from family member in lieu of salivary cotinine verification. At Month 12, salivary cotinine will be used for biochemical validation of all smokers reporting abstinence.
number of 24-hour quit attempts (smoker participants) | 12 months
  self-report of making quit attempts that lasted at least for 24 hours since baseline
use of smoking cessation resources since program initiation (smoker participants) | 12 months
  Use of evidence-based smoking cessation resources since program initiation
at least 50% reduction of the amount of cigarettes smoked per day from baseline | 12 months
  smoking reduction

CONTACTS AND LOCATIONS:
Overall Officials: Janice Y Tsoh, PhD, Principal Investigator — University of California, San Francisco
Locations (3):
- United States (3):
  - Southeast Asian Community Center (SEACC), San Francisco, California
  - Chinese Community Health Resource Center, San Francisco, California
  - Vietnamese Voluntary Foundation, San Jose, California